CLINICAL TRIAL: NCT01642927
Title: Pulse Wave Analysis in Advanced Heart Failure Patients Before and After Ventricular Assist Device
Brief Title: Pulse Wave Analysis in Advanced Heart Failure
Acronym: PWA-HF
Status: Withdrawn | Type: Observational
Why Stopped: PI left University
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: FWA00000312-7
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Left Ventricular Assist Device; Heart Failure; Intra-aortic Balloon Pump; LVAD Clot; LVAD-related GI Bleed
Keywords: LVAD; IABP; Heart Failure; Thrombosis; Hemorrhage
MeSH Terms: conditions — Heart Failure; Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Intra-Aortic Balloon Pump (IABP) Group: Advanced Heart Failure and/or pre-LVAD surgical patient with IABP
- IABP/LVAD Group: Post-LVAD surgical patients with IABP
- Post-LVAD Group: LVAD patients 3 months or greater post-implantation undergoing echocardiography
- LVAD Event Group: LVAD patients who have developed LVAD thrombosis or GI hemorrhage related to LVAD
- Arrhythmia group: LVAD patient with an irregular heartbeat.
- Valvular disease group: LVAD patient with valvular heart disease
- Normal control group: Healthy participant without any known heart disease (Control group).

SUMMARY:
A comparison of pulse wave characteristics, as measured by peripheral tonometry, in pre and post Left Ventricular Assist Device (LVAD) patients.

DETAILED DESCRIPTION:
Pulse waveforms, especially central pressure waveforms, are predictive of cardiovascular events. Peripheral waveforms have been correlated to central waveforms. Peripheral waveforms can be easily measured through applanation tonometry. In this study the investigators hypothesize:

1. That previously established peripheral tonometry techniques would apply to patients with advanced heart failure, including continuous flow LVADs and facilitate serial evaluation of central hemodynamics without invasive monitoring.
2. That temporary changes in LVAD speed will be evident in frequency spectrum analysis of peripheral, non-invasive waveforms.
3. That clinical events involving LVAD will have characteristic frequency spectra.

ELIGIBILITY:
Inclusion Criteria:

1)18 years of age or older

2)Advanced heart failure as defined by need for IABP or LVAD

3)One or more of the following:

* Current inpatient heart failure treatment with intra-aortic balloon pump (IABP)-IABP Group

  •≤ 1 week post-LVAD implantation with current IABP support-IABP/LVAD Group

  •≥ 3 mo post-LVAD placement and scheduled for LVAD speed optimization with echocardiography.-Post-LVAD Group
* Post-LVAD placement with suspected GI hemorrhage or LVAD thrombosis-LVAD Event Group

  4)Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. Clinical status will not permit pause of IABP (IABP and IABP/LVAD Groups)
2. Unable to undergo echo or oversewn or patched aortic valve (Post-LVAD Group)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced heart failure patients, eligible for or currently treated with LVAD, outpatient cardiology clinic or inpatient heart failure service patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Observation of pulse wave signatures in LVAD patients | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eckman, MD, Principal Investigator — University of Minnesota
Locations (1):
- Univeristy of Minnesota Lillehei Heart Institute, Minneapolis, Minnesota, United States